CLINICAL TRIAL: NCT00729573
Title: Phase 2B Safety and Effectiveness Study of Tenofovir 1% Gel, Tenofovir Disproxil Fumarate Tablet and Emtricitabine/Tenofovir Disoproxil Fumarate Tablet for the Prevention of HIV Infection in Women
Brief Title: Bone Mineral Density Substudy - An Ancillary Study to MTN-003
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Microbicide Trials Network (Network)
Responsible Party: Sponsor
Other Study IDs: MTN-003B; 10709 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV Seronegativity; Bone Mineral Density
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples

GROUPS / COHORTS (1):
- 1: Participants in MTN-003. Participants will remain a part of their assigned MTN-003 study groups.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Emtricitabine/tenofovir disoproxil fumarate placebo; Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate placebo

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil fumarate — 200 mg/300 mg tabletas a part of MTN-003
  Other Names: FTC/TDF; Truvada
Drug: Emtricitabine/tenofovir disoproxil fumarate placebo — placebo tablet as a part of MTN-003
  Other Names: FTC/TDF placebo; Truvada placebo
Drug: Tenofovir disoproxil fumarate — 300 mg tablet as a part of MTN-003
  Other Names: TDF
Drug: Tenofovir disoproxil fumarate placebo — placebo tablet as a part of MTN-003
  Other Names: TDF placebo

SUMMARY:
The MTN-003 HIV prevention study include the use of microbicides, substances that kill microbes, and tenofovir disoproxil fumarate (TDF) and emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) - oral, FDA-approved, anti-HIV drugs. The purpose of this study is to determine if taking daily TDF and FTC/TDF as a part of the study MTN-003 has an effect on bone mineral density (BMD).

DETAILED DESCRIPTION:
The effect of tenofovir on bone mineral density (BMD) has not yet been studied and is of potential concern. The purpose of this study is to determine the changes in BMD among individuals receiving TDF and FTC/TDF compared with a placebo.

This substudy will enroll individuals currently participating in MTN-003. The expected duration of participation for each participant is approximately 48 months. Study treatment will be provided by MTN-003. Study treatment will not be provided by this substudy.

Study visits will occur every 6 months after enrollment. A nutrition assessment, physical activity history, and urine and blood collection will occur at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in MTN-003
* Randomized to oral study product in MTN-003 within 14 days prior to study entry

Exclusion Criteria:

* Medical condition known to affect bone or taking any medication known to affect bone. More information on this criterion can be found in the protocol.
* Permanently discontinued from oral study product in MTN-003 prior to study entry
* Any condition that, in the opinion of the investigator, would interfere with the study
* Pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sexually active, HIV-uninfected women who are currently enrolled in MTN-003
Sampling Method: Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density | Throughout study

SECONDARY OUTCOMES:
Changes in nutrition | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Riddler, MD, MPH, Study Chair — University of Pittsburgh
Locations (4):
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Zimbabwe (3):
  - Seke South CRS, Chitungwiza
  - Zengeza CRS, Chitungwiza
  - Spilhaus CRS, Harare

REFERENCES:
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Background] Rosen RK, Morrow KM, Carballo-Dieguez A, Mantell JE, Hoffman S, Gai F, Maslankowski L, El-Sadr WM, Mayer KH. Acceptability of tenofovir gel as a vaginal microbicide among women in a phase I trial: a mixed-methods study. J Womens Health (Larchmt). 2008 Apr;17(3):383-92. doi: 10.1089/jwh.2006.0325. PMID 18328009